CLINICAL TRIAL: NCT05597540
Title: Efficacy of 7 Days Versus 14 Days of Antibiotic Therapy for Acute Pyelonephritis in Kidney Transplant Recipients, a Multicentre Randomized Non-inferiority Trial.
Acronym: SHORTCUT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP200020
Record Dates: First submitted 2022-10-24; First posted 2022-10-28 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-02

CONDITIONS: Pyelonephritis Acute; Kidney Transplant Infection
Keywords: antibiotic therapy; duration of antibiotic treatment reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Randomized double blind trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 7 day-duration antibiotic treatment (Experimental)
  Interventions: Drug: Short antibiotic treatment
- 14 day-duration antibiotic treatment (Active Comparator)
  Interventions: Drug: Usual antibiotic treatment

INTERVENTIONS:
Drug: Short antibiotic treatment — 7 day-duration antibiotic treatment. The choice of antibiotic treatment is left to the medical team in charge of the patient.
  Arms: 7 day-duration antibiotic treatment
Drug: Usual antibiotic treatment — 14 day-duration antibiotic treatment. The choice of antibiotic treatment is left to the medical team in charge of the patient.
  Arms: 14 day-duration antibiotic treatment

SUMMARY:
Infections are a major cause of morbidity and mortality in solid organ transplant recipients. In kidney transplant recipients (KTR) urinary tract infection (UTI) represent 45-72% of all infections, and 30% of all hospitalizations for sepsis. Acute transplant pyelonephritis are the most common complications occurring in more than 20% of patients, mainly in the first year after transplantation. They are associated with an increased risk of acute kidney rejection and long-term kidney graft dysfunction. Gram-negative bacteria, mainly E. coli, account for more than 70% of UTI in KTR. As those infections are favoured by urinary tract modifications/defects and immunosuppression, they are often recurrent and necessitate repeated courses of antibiotics. Selective pressure due to antibiotic consumption, along with frequent hospital admissions and immunosuppression, are well known risk factors for the development of antibiotic resistant infections. Multidrug (MDR)- or extensively (XDR)- drug resistant Enterobacteriaceae including ESBL- or carbapenemase-producing organisms, are thus increasingly observed in transplant units and represent a global threat as very few new antibiotics are expected in the next decade.

One main strategy to limit antimicrobial resistance is to reduce the duration of antibiotic treatment. A 7 day-course is recommended for simple acute pyelonephritis (APN) treated with fluoroquinolones or parenteral B-lactams, prolonged up to 10 or 14 days in the presence of underlying disease at risk of complications. Most KT teams treat patients between 14-21 days as recommended by American guidelines. However, the need to extend treatment duration in immunosuppressed patients is a poorly defined concept and the optimal duration of treatment for APN in KTR is not known as these patients are excluded from most studies.

As there is an urgent need to reduce antibiotic consumption in this population at high risk of developing infections due to resistant pathogens, the hypothesis is that a 7 day-treatment is sufficient to cure APN with good clinical response after 48h of treatment in KTR and is as effective as 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years KTR
* APN defined by: fever (T°≥38°C) (with or without clinical signs and/or symptoms of UTI) and pyuria (≥10^4 white blood cells/mL or ≥10/mm3) and positive urine culture (uropathogen ≥10^3 CFU/mL susceptible to the empirically administrated antibiotic)
* No confirmed or suspected febrile non urinary bacterial infection
* No urologic/renal complication at baseline imaging (abscess, obstruction...)
* Favourable early response to antibiotic treatment:48 to 60 hours after the first dose of antibiotic effective against the causative uropathogen) defined by: T°<38°C and improvement (or resolution) of signs and/or symptoms of urinary tract infection if present at diagnosis
* Written informed consent

Exclusion Criteria:

* Severe or complicated condition

  * Any rapidly progressing disease or immediately life-threatening illness, including, but not limited to, septic shock, current or impeding respiratory failure, acute heart or liver failure
  * Admission or stay in intensive care unit at baseline
  * Obstruction of the urinary tract
  * Renal, perinephric or prostatic abscess
* Prior inclusion in this study
* Current participation to another interventional study
* Dual antibiotic therapy (prophylactic antibiotic such as cotrimoxazole allowed) (only 1 dose of aminoside is allowed before randomization)
* First month post transplantation
* Current indwelling catheter (including bladder catheter, ureteral stents, percutaneous nephrostomy tubes)
* Neurogenic bladder
* Enterocystoplasty
* Immunodeficiency or immunosuppressive therapy not related to kidney transplantation including hematologic malignancy, cancer, asplenia, neutropenia<500 neutrophils/mm3
* Pregnancy, breastfeeding
* Hypersensitivity or previous severe adverse drug reaction to the antibiotic therapy
* Unable or unwilling, in the judgment of the investigator, to comply with the protocol
* Life expectancy<1 month
* Patient under legal guardianship or without healthcare coverage
* Homeless patient
* Women with childbearing potential not using adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2027-03-22 (Estimated); Study Completion 2027-08-22 (Estimated)

PRIMARY OUTCOMES:
Clinical cure day 30 | at day 30
  Clinical cure and no additional antibiotic treatment since the end of antibiotic treatment up to the main evaluation at day 30.
  Clinical cure is defined as fever <38°C and no symptoms of Urinary Tract Infection (UTI).

SECONDARY OUTCOMES:
Clinical cure day 90 | at day 90
  Clinical cure and no additional antibiotic treatment since the end of antibiotic treatment up to the main evaluation at day 90.
  Clinical cure is defined as fever <38°C and no symptoms of Urinary Tract Infection (UTI).
Clinical cure day 180 | at day 180
  Clinical cure and no additional antibiotic treatment since the end of antibiotic treatment up to the main evaluation at day 180.
  Clinical cure is defined as fever <38°C and no symptoms of Urinary Tract Infection (UTI).
Microbiological cure day 30 | at day 30
  Microbiological cure is defined as a sterile urine or uropathogene ≤ 10.3 CFU/mL in urine culture
Microbiological cure day 90 | at day 90
  Microbiological cure is defined as a sterile urine or uropathogene ≤ 10.3 CFU/mL in urine culture
Microbiological cure day 180 | at day 180
  Microbiological cure is defined as a sterile urine or uropathogene ≤ 10.3 CFU/mL in urine culture
Incidence of relapse/recurrence day 30 | at day 30
  Relapse or recurrence of the Urinary Tract Infection
Incidence of relapse/recurrence day 90 | at day 90
  Relapse or recurrence of the Urinary Tract Infection
Incidence of adverse event | at day 180
  Incidence of adverse events imputable to antibiotic treatment
Kidney function | at day 90
  Evaluated by MDRD or CKD
  MDRD : Modification of Diet in Renal Disease (MDRD) Study equation.
  Froissart M, Rossert J, Jacquot C, Paillard M, Houillier P. Predictive performance of the modification of diet in renal disease and Cockcroft-Gault equations for estimating renal function. J Am Soc Nephrol 2005;16(3):763-73.
  CKD-EPI (Chronic Kidney Disease EPIdemiology collaboration, Levey, 2009)
  A New Equation to Estimate Glomerular Filtration Rate. Andrew S. Levey, MD; Lesley A. Stevens, MD, MS; Christopher H. Schmid, PhD; Yaping (Lucy) Zhang, MS; Alejandro F. Castro III, MPH; Harold I. Feldman, MD, MSCE; John W. Kusek, PhD; Paul Eggers, PhD; Frederick Van Lente, PhD; Tom Greene, PhD; and Josef Coresh, MD, PhD, MHS, for the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration). Annals of Internal Medicine 2009;150(9):604-613
Kidney function | at day 180
  Evaluated by MDRD or CKD
  MDRD : Modification of Diet in Renal Disease (MDRD) Study equation.
  Froissart M, Rossert J, Jacquot C, Paillard M, Houillier P. Predictive performance of the modification of diet in renal disease and Cockcroft-Gault equations for estimating renal function. J Am Soc Nephrol 2005;16(3):763-73.
  CKD-EPI (Chronic Kidney Disease EPIdemiology collaboration, Levey, 2009)
  A New Equation to Estimate Glomerular Filtration Rate. Andrew S. Levey, MD; Lesley A. Stevens, MD, MS; Christopher H. Schmid, PhD; Yaping (Lucy) Zhang, MS; Alejandro F. Castro III, MPH; Harold I. Feldman, MD, MSCE; John W. Kusek, PhD; Paul Eggers, PhD; Frederick Van Lente, PhD; Tom Greene, PhD; and Josef Coresh, MD, PhD, MHS, for the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration). Annals of Internal Medicine 2009;150(9):604-613
Hospital length of stay | Up to day 180
  Hospitalisation length stay defined by the delay between the date of inclusion and the date of hospital discharge
Antibiotic consumption | Up to day 180
  Antibiotic consumption (indication, dose and duration) throughout the follow-up will be recorded.
Rectal carriage | at inclusion
  Rectal carriage of antibiotic resistant Enterobacteriaceae
Rectal carriage | at day 30
  Rectal carriage of antibiotic resistant Enterobacteriaceae

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - CHU Bordeaux, Bordeaux
  - Hôpital Foch, Boulogne-Billancourt
  - CHU Mondor, Créteil
  - CHU Lyon, Lyon
  - CHU Nantes, Nantes
  - CHU Kremlin-Bicêtre, Paris
  - CHU Necker, Paris
  - CHU Saint Louis, Paris
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided